CLINICAL TRIAL: NCT06447532
Title: Use of Machine Learning Techniques for Serial Assessment of Systemic Inflammatory Markers in Breast Cancer Patients
Acronym: INFLAMMATE
Status: Enrolling by invitation | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Collaborators: Kansai Medical University (Other); University of Sao Paulo (Other); Kyoto University (Other); Barretos Cancer Hospital (Other); Women's College Hospital (Other); Emory University (Other); University of Campinas, Brazil (Other); Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other); Instituto Nacional de Cancer, Brazil (Other Government); Universidade Federal do Triangulo Mineiro (Other); Instituto de Cardiología y Medicina Vascular Hospital Zambrano-Hellion Tec Salud (Other); Hospital Vall d'Hebron (Other); Mansoura University (Other); Seoul National University (Other)
Responsible Party: Principal Investigator, Afonso Celso Pinto Nazario, Professor and Coordinator at the Department of Gynecology at EPM/UNIFESP., Federal University of São Paulo
Other Study IDs: University of Sao Paulo
Record Dates: First submitted 2024-04-26; First posted 2024-06-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; machine learning; prognosis; inflammation
MeSH Terms: conditions — Breast Neoplasms; Inflammation | interventions — Surgical Procedures, Operative; Mastectomy; Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group I: Breast cancer: All the participants involved in our study are women who are diagnosed breast cancer and treated with surgery or neoadjuvant chemotherapy from January 1st 2013 to December 31st 2018.
  Interventions: Procedure: Surgery (Mastectomy or quadrantectomy)

INTERVENTIONS:
Procedure: Surgery (Mastectomy or quadrantectomy) — Surgery (mastectomy or quadrantectomy); Neoadjuvant chemotherapy
  Other Names: Neoadjuvant chemotherapy

SUMMARY:
Breast cancer is the most common cancer in women globally, with 2.3 million new cases diagnosed in 2020. Hormone receptor positive (HR+), human epidermal growth factor receptor 2 negative (HER2-) breast cancer is the most prevalent subtype, comprising 69% of all breast cancers in the USA. Within the tumor immune microenvironment, a higher intensity of myeloid cell infiltration and low levels of lymphocyte infiltration have been associated with worse outcomes. Markers in peripheral blood have emerged as predictive biomarkers that can be easily obtained non-invasively and at low cost. Experiments have confirmed the relative components of these tests (such as the immune cells) directly or indirectly participated in tumour occurrence, development, and immune escape, underscoring the potential use of laboratory tests as tumour biomarkers

DETAILED DESCRIPTION:
In breast cancer, increased neutrophil levels and decreased lymphocyte levels in peripheral blood are associated with worse overall survival (OS). In HR+, HER2- metastatic breast cancers, low pretreatment NLR and high pretreatment absolute lymphocyte count (ALC) were related with better progression-free survival (PFS) and OS. The development of predictive models, based on machine learning (ML) algorithms it has been used in prognostication and assist in the diagnosis of different types of cancer.

Although regular laboratory tests have potential to be breast cancer biomarkers, a single test is yet to provide adequate sensitivity or specificity. Artificial intelligence (AI) could help with integrating data from multiple tests to aid diagnosis. Technical improvements such as data storage capacity, computing power, and better algorithms mean that ML can process clinically meaningful information from laboratory test data. Models' generalisability and stability still need to be confirmed, in view of limitations such as the absence of various pathological types, small cohorts, and lack of external validation. Therefore, a competitive model is also essential to achieve more accurate stratification of patients with breast cancer. The purpose of this retrospective multicentre study is to systematically evaluate the ability of laboratory tests to predict breast cancer, and develop a robust and generalisable model to assist in identifying patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women patients with age between 18 and 75 years old;
* Invasive breast carcinoma patients diagnosed by pathology ;
* Patients diagnosed between 1 January 2013 and 31 December 2018;
* Have a complete blood count performed before the surgical intervention (mastectomy or conservative breast surgery) or neoadjuvant chemotherapy;

Exclusion Criteria:

Presence of hematological disorders;

* Bilateral breast cancer;
* Male;
* Karnofsky Performance Status Score < 70';
* Inflammatory breast cancer and in situ carcinoma;
* Pregnancy or breastfeeding;
* Evidence of local or distant recurrence.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women diagnosed with breast cancer.
Study Population: All the women involved in our study are patients who are diagnosed breast cancer pathologically and treated with surgery or neoadjuvant chemotherapy from January 1st 2013 to December 31st 2018.
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the date of diagnosis to the date of death, assessed up to 120 months
  Overall survival

SECONDARY OUTCOMES:
Disease free survival | From the date of diagnosis to the date of first progression (local recurrence of tumor or distant metastasis), assessed up to 60 months
  Disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Afonso C Nazario, PhD, Principal Investigator — University Federal of Sao Paulo
Locations (13):
- Pablo Mandó, Buenos Aires, Buenos Aires, Argentina
- Brazil (5):
  - Rosekeila Simoes Nomeline, Uberaba, Minas Gerais
  - Tomás Reinert, Porto Alegre, Rio Grande do Sul
  - Idam Oliveira Junior, Barretos, São Paulo
  - César Cabello, Campinas, São Paulo
  - Daniel Guimaraes Tiezzi, Ribeirão Preto, São Paulo
- Vasily Giannakeas, Toronto, Ontario, Canada
- Salma Elashwah, Cairo, Egypt
- Japan (2):
  - Masahiro Takada, Osaka, Osaka
  - Masakazu Toi, Tokyo, Tokyo
- Cynthia Mayte Villarreal Garza, Mexico City, Mexico
- Wonshik Han, Seoul, South Korea
- Cristina Saura, Madrid, Spain, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Faria SS, Giannarelli D, Cordeiro de Lima VC, Anwar SL, Casadei C, De Giorgi U, Madonna G, Ascierto PA, Mendoza Lopez RV, Chammas R, Capone M. Development of a Prognostic Model for Early Breast Cancer Integrating Neutrophil to Lymphocyte Ratio and Clinical-Pathological Characteristics. Oncologist. 2024 Apr 4;29(4):e447-e454. doi: 10.1093/oncolo/oyad303. PMID 37971409
- [Background] Choi E, Bahadori MT, Schuetz A, Stewart WF, Sun J. Doctor AI: Predicting Clinical Events via Recurrent Neural Networks. JMLR Workshop Conf Proc. 2016 Aug;56:301-318. Epub 2016 Dec 10. PMID 28286600